CLINICAL TRIAL: NCT05826054
Title: Phase 1 Dose Escalating Study for Montbretin a
Brief Title: Montbretin Clinical Trial in Healthy Volunteers and Type 2 Diabetics
Acronym: MbA
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Robert Petrella (Other)
Collaborators: Michael Smith Foundation for Health Research (Other); Canadian Glycomics Network (GlycoNet) - Networks of Centres of Excellence (NCE) (Unknown)
Responsible Party: Sponsor-Investigator, Robert Petrella, Professor and Head (Chair), Department of Family Practice, University of British Columbia
Organization: University of British Columbia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MbA01
Record Dates: First submitted 2023-04-11; First posted 2023-04-24 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; Montbretin A; Type II Diabetes Mellitus Without Complication; Noninsulin-Dependent Diabetes Mellitus; Healthy participants
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — montbretin A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): In this study, participants will receive increasing dosages of the Study Treatment (Montbretin A, MbA) at each treatment visit. The Study Treatment will be taken with a standardized meal (a meal that has specified quantities of carbohydrates, fats and proteins). At each visit, participants will receive one dose (in pill form) of MbA. As long as they are not experiencing any side effects, this dose will be gradually increased at each study visit (starting from 10 mg, 25 mg, 50 mg, 100 mg, 200 mg, to 300 mg MbA).
  Interventions: Dietary Supplement: Montbretin A

INTERVENTIONS:
Dietary Supplement: Montbretin A — The investigational product is 95% pure montbretin A (MbA), a glycosylated acyl-flavonol isolated from the corms (bulbs) of the Crocosmia plant through hot water extraction. It is a potent and specific inhibitor of human pancreatic amylase (HPA).

SUMMARY:
The goal of this clinical trial is to test the investigational product, Montbretin A (MbA) in either individuals with type 2 diabetes (T2D) or healthy participants.

The main questions it aims to answer are:

* Safety of MbA
* Whether MbA has less side effects in comparison to other medications used to treat T2D

Participants will:

* Be given MbA at increasing amounts (10 mg to 300 mg) over a two-week treatment period, along with standardized meal;
* Undergo testing, including blood draws, blood sugar checks, electrocardiogram (ECG) and questionnaires.

DETAILED DESCRIPTION:
BACKGROUND: Diabetes is an increasingly common disease that affects 6% of the population. It is a chronic metabolic disorder because the body cannot produce enough insulin or cannot respond well to insulin to control the amount of sugar in the blood. Insulin is a hormone secreted by the pancreas that increases the ability of tissues to absorb blood glucose. After a meal, our body will break down the nutrients in the food we eat, such as carbohydrates. These smaller nutrients are then absorbed in our small intestine into our blood. Without proper insulin function, our body is unable to lower the blood sugar and use the blood sugar correctly, leading to high blood sugar (also known as hyperglycemia). Over time, this can lead to complications in the eyes, nervous system, kidney and heart.

One type of diabetes medications, alpha-glucosidase inhibitors (AGIs), prevent blood sugar spikes (period of out of control high blood sugar levels) in diabetic patients after a meal. This type of medication prevents breakdown of carbohydrates into small sugars that can be absorbed in the gut. AGIs usually work well in preventing blood sugar spikes, but they have a number of side effects such as increased gas, bloating and diarrhea. Because of this, patients usually do not follow the recommended schedule for taking AGIs, which means the medications wont work as well.

The Study Treatment ("Montbretin A") provides another way to control blood sugar spikes after a meal. This method targets an enzyme (substance produced by body to help break down substances) found in the small intestine called human pancreatic amylase (HPA), which helps in the first step of breaking down carbohydrates. The Study Treatment works by blocking HPA from performing its function. This could potentially be used to treat T2D by preventing the initial breakdown of carbohydrates, which can lead to less sugars absorbed to the blood and better blood sugar control. MbA will lead to larger pieces of carbohydrates passed to the colon, reducing the speed of gas produced. This might lead to reduced stomach upsets.

MAIN AIM: To test the safety and tolerability (in terms of stomach-related side effects) of MbA in humans.

METHOD: This is an open-label, first-in-human, single-arm, single-center Phase I clinical trial. Participants will receive increasing dose of MbA (starting from 10 mg to 300 mg) with a standardized meal during the two-week treatment period (Weeks 1 and 2), with follow-up visits scheduled in Week 3 (one week after treatment completion) and Week 12 (nine weeks after treatment completion).

Participants are expected to participate for up to 13 weeks. This include one screening visit (one week prior to start of treatment), 2 weeks of treatment (3 visits per week for a total of 6 visits), and 2 follow-up visits (one week and nine weeks after completing treatment).

The tests that will be done in this study include:

* One blood draw at each visit
* Electrocardiogram (ECG), at screening and the first follow up visit
* Blood sugar checks, including one finger prick and continuous glucose monitoring using a device at screening and each treatment visit
* Questionnaire regarding gastrointestinal symptoms
* Gastro-Intestinal Diary (GID), which needs to be filled in daily after screening and up to one week after treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age ≤ 65 years; ≥19 years;
* Have diagnosed type-2 diabetes mellitus with HbA1C between 6.5% to 11% that is currently managed by diet and no other medications or healthy volunteers defined as not having diagnosis of type-2 diabetes mellitus.
* Have routine and normal dietary habits that include three meals a day;
* Normal hematological parameters as determined through an in-person screening blood draw including HbA1C >4.0% in healthy volunteers.
* Use of an effective barrier method of birth control throughout the study, surgical sterility, or menopausal for at least 2 years;
* In the study team's opinion, capable of understanding the visit schedule requirement and study medication dosing requirements.
* Be able to avoid all supplements that affect blood sugar for the duration of the study eg. chromium, bitter melon, thiamine, berberine, alpha-lipoic acid, devil's claw, horse chestnut, fenugreek, ginseng, psyllium, cinnamon, garlic and panax.

Exclusion Criteria:

* Currently in poor health, as determined by the study doctor
* Currently on medication, except vitamins and/or birth control
* Not eating three regular meals a day
* Current or a history of impairment of gastro-intestinal function, including but not limited to inflammatory bowel disease, colonic ulceration, and/or partial intestinal obstruction
* Travelled to a foreign country less than four (4) weeks prior to study entry;
* Surgery less than four (4) weeks a prior to study entry;
* Pregnant or lactating women;
* Planning to participate in other investigational drugs while participating in the study;
* Known allergy to study medication or its components (non-medicinal ingredients); and
* A history of noncompliance to medical regimens or inability or unwillingness to return for all scheduled visits

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 2 weeks
  The MTD is defined as the minimum dose that results in a dose limiting toxicity in the form of gastro-intestinal adverse events (relevant flatulence and/or diarrhea as determined by the Gastrointestinal Symptom Rating Scale) in 33% of the test subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Petrella, MD, PhD, Principal Investigator — University of British Columbia
Locations (1):
- VCHRI Clinical Research Unit, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No